CLINICAL TRIAL: NCT02510742
Title: Physiological Changes Induced With SPG Stimulation in Migraine Patients - Amendment to the Pathway M-1 Trial
Brief Title: Physiological Changes With SPG Stimulation in Migraine Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Song Guo, MD, PhD student, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H-1-2011-152
Record Dates: First submitted 2015-07-22; First posted 2015-07-29 (Estimated); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Chronic Migraine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- SPG neurostimulation (Active Comparator): SPG neurostimulation of frequency 20 Hz
  Interventions: Device: Neurostimulation
- Control (Sham Comparator): Sham neurostimulation of amplitude=0
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Neurostimulation — Neurostimulation of sphenopalatine ganglion (SPG) of 20 Hz
  Arms: SPG neurostimulation
Device: Sham stimulation — Sham stimulation of sphenopalatine ganglion (SPG) with amplitude=0
  Arms: Control

SUMMARY:
Hypothesis:

Stimulation of the SPG at low frequencies (20 Hz)is believed to cause a physiological parasympathetic upregulation which increases VMCA, concentration and cephalic vessel diameter.

ELIGIBILITY:
Inclusion Criteria:

* Chronic migraine patients

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-07; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Changes of mean blood velocity of middle cerebral artery (VMCA) using transcranial Doppler upon low frequency SPG stimulation | 0-90 min

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Headache Center, Copenhagen, Glostrup, Denmark

REFERENCES:
- [Derived] Guo S, Falkenberg K, Schytz HW, Caparso A, Jensen RH, Ashina M. Low frequency activation of the sphenopalatine ganglion does not induce migraine-like attacks in migraine patients. Cephalalgia. 2020 Aug;40(9):966-977. doi: 10.1177/0333102420921156. Epub 2020 Apr 22. PMID 32321288